CLINICAL TRIAL: NCT07294456
Title: Evaluation of Periodontal Status in Individuals With Hidradenitis Suppurativa: A Cross-Sectional Study
Brief Title: Periodontal Status and Disease Severity in Hidradenitis Suppurativa Patients
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Şeyma Çardakçı, ASSİSTANT PROFESSOR, Saglik Bilimleri Universitesi
Other Study IDs: SUDE1824
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: HİDRADENİTİS SUPPURATİVA
Keywords: HİDRADENİTİS SUPPURATİVA; PERİODONTAL DİSEASE; PERİODONTİTİS; GİNGİVAL İNFLAMMATİON
MeSH Terms: conditions — Hidradenitis Suppurativa; Gingival Diseases; Dry Socket; Gingivitis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hidradenitis Suppurativa Group: Participants diagnosed with hidradenitis suppurativa undergoing periodontal examination.
  Interventions: Other: No intervention (observational study)
- Healthy Control Group: Systemically healthy individuals without hidradenitis suppurativa undergoing periodontal examination.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — Observational study with no treatment or intervention applied.

SUMMARY:
This cross-sectional study aims to evaluate the periodontal status of individuals diagnosed with hidradenitis suppurativa (HS) and to compare them with systemically healthy controls. HS is a chronic inflammatory skin disease characterized by recurrent lesions and systemic inflammation, which may influence periodontal health. In this study, periodontal parameters-including probing depth, clinical attachment loss, gingival index, plaque index, and bleeding on probing-will be assessed using standard clinical methods. Dermatological examination will include disease duration, lesion characteristics, and Hurley staging. The study will investigate the prevalence of periodontitis in HS patients and explore potential associations between periodontal findings and HS severity. Findings from this research may provide insight into shared inflammatory pathways and contribute to understanding the possible link between HS and periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of hidradenitis suppurativa.
* Age greater than 18 years.
* Presence of at least 12 teeth in the mouth, excluding third molars.

Exclusion Criteria:

* Age under 18 years.
* Pregnancy.
* Breastfeeding.
* Receiving treatment for periodontitis or hidradenitis suppurativa within the past 3 months.
* Use of antibiotics, anti-inflammatory drugs, or immunomodulatory medications within the past 3 months.

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult individuals with a confirmed diagnosis of hidradenitis suppurativa and age-matched healthy controls, each having at least 12 teeth (excluding third molars), and no recent periodontal or systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Correlation Between Periodontal Status and Hidradenitis suppurativa | Baseline (single assessment)

SECONDARY OUTCOMES:
Correlation between Periodontal Status and Hurley Stage | Baeline (single assesment)
Corralation between Hurley Stage and Oral Health Impact Profile OHIP-14) Score | baseline (single assesment)
Correlation between Dermatology Life Quality Index (DLQI) and Oral Health Impact Profile (OHIP-14) Total Score | baseline (single assesment)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gülhane Faculty of Dentistry, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided